CLINICAL TRIAL: NCT00002654
Title: Phase III Study of Hyperfractionated Radiation Therapy With or Without Simultaneaous Application of CIS-Platinum in Patients With Moderately Advanced to Advanced Cancers of the Head and Neck
Brief Title: Radiation Therapy With or Without Cisplatin in Treating Patients With Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: SAKK 10/94; SWS-SAKK-10/94; EU-94039; CDR0000064188
Record Dates: First submitted 1999-11-01; First posted 2004-07-01 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Drug Therapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: chemotherapy
Drug: cisplatin
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if radiation therapy plus chemotherapy is more effective than radiation therapy alone in treating patients with advanced head and neck cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy plus cisplatin with radiation therapy alone in treating patients with advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the time to treatment failure (local and regional) in patients with moderately advanced and advanced squamous cell carcinoma of the head and neck (no distant metastases) when treated with hyperfractionated radiotherapy with vs. without 2 courses of simultaneously administered cisplatin. II. Assess the time to distant metastatic relapse, overall survival, and toxicity in patients receiving these treatments. III. Evaluate whether the potential tumor-doubling time is an indicator for risk of treatment failure in patients receiving these treatments.

OUTLINE: Randomized study. Arm I: Radiotherapy plus Single-Agent Chemotherapy followed, as indicated, by Surgery. Hyperfractionated external-beam tumor irradiation using photon energies of 4-6 MV or electrons of 6-12 MV (interstitial brachytherapy boost to lesions of the oral cavity allowed); plus Cisplatin, CDDP, NSC-119875; followed, in patients with persistent disease (at the discretion of the surgeon), by resection of primary tumor or involved nodes. Arm II: Hyperfractionated radiotherapy followed by Surgery. Tumor irradiation as in Arm I; followed by resection as in Arm I.

PROJECTED ACCRUAL: At least 400 patients will be accrued over 5 years. Interim analyses to allow for early stopping will be carried out after entry of 50 and 100 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically documented squamous cell cancer of the head and neck in the following sites: Hypopharynx Larynx Oral cavity Oropharynx Stage III/IV disease No distant metastases by the following: Chest x-ray (all patients) Liver ultrasound or CT and bone scintigraphy (all hypopharyngeal cancers, those with involved lower neck nodes, and as clinically indicated) Multiple sites of disease eligible provided radiotherapy treatment volume remains acceptable

PATIENT CHARACTERISTICS: Age: 20 to 75 Performance status: WHO 0-2 Hematopoietic: WBC greater than 3,000 Platelets greater than 100,000 Hepatic: Not specified Renal: Creatinine clearance at least 60 ml/min No renal disease or impairment of renal function Cardiovascular: No coronary heart disease No cardiac failure No history of pulmonary embolism within 2 years Other: No clinical hearing impairment No peripheral neuropathy with concomitant handicap No severe diabetes mellitus with serious vasculopathy or neuropathy No second cancer except: Nonmelanomatous skin or lip cancer In situ carcinoma of the cervix Blood/body fluid analyses to determine eligibility completed within 14 days prior to registration

PRIOR CONCURRENT THERAPY: No prior treatment for head and neck cancer Excisional biopsy for diagnosis allowed

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 1994-04; Primary Completion 1999-03 (Actual); Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pia Huguenin, MD, Study Chair — UniversitaetsSpital Zuerich
Locations (1):
- Universitaetsspital, Zurich, Switzerland

REFERENCES:
- [Result] Ghadjar P, Simcock M, Studer G, Allal AS, Ozsahin M, Bernier J, Topfer M, Zimmermann F, Betz M, Glanzmann C, Aebersold DM; Swiss Group for Clinical Cancer Research (SAKK). Concomitant cisplatin and hyperfractionated radiotherapy in locally advanced head and neck cancer: 10-year follow-up of a randomized phase III trial (SAKK 10/94). Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):524-31. doi: 10.1016/j.ijrobp.2010.11.067. Epub 2011 Feb 16. PMID 21300466
- [Result] Taussky D, Rufibach K, Huguenin P, Allal AS. Risk factors for developing a second upper aerodigestive cancer after radiotherapy with or without chemotherapy in patients with head-and-neck cancers: an exploratory outcomes analysis. Int J Radiat Oncol Biol Phys. 2005 Jul 1;62(3):684-9. doi: 10.1016/j.ijrobp.2004.11.027. PMID 15936546
- [Result] Huguenin P, Beer KT, Allal A, Rufibach K, Friedli C, Davis JB, Pestalozzi B, Schmid S, Thoni A, Ozsahin M, Bernier J, Topfer M, Kann R, Meier UR, Thum P, Bieri S, Notter M, Lombriser N, Glanzmann C. Concomitant cisplatin significantly improves locoregional control in advanced head and neck cancers treated with hyperfractionated radiotherapy. J Clin Oncol. 2004 Dec 1;22(23):4665-73. doi: 10.1200/JCO.2004.12.193. Epub 2004 Nov 8. PMID 15534360
- [Result] Ghadjar P, Simcock M, Zimmermann F, Betz M, Bodis S, Bernier J, Studer G, Aebersold DM; Swiss Group for Clinical Cancer Research (SAKK). Predictors of severe late radiotherapy-related toxicity after hyperfractionated radiotherapy with or without concomitant cisplatin in locally advanced head and neck cancer. Secondary retrospective analysis of a randomized phase III trial (SAKK 10/94). Radiother Oncol. 2012 Aug;104(2):213-8. doi: 10.1016/j.radonc.2012.05.004. Epub 2012 Jun 21. PMID 22726581
- [Result] Ghadjar P, Pottgen C, Joos D, Hayoz S, Baumann M, Bodis S, Budach W, Studer G, Stromberger C, Zimmermann F, Kaul D, Plasswilm L, Olze H, Bernier J, Wust P, Aebersold DM, Budach V. Haemoglobin and creatinine values as prognostic factors for outcome of concurrent radiochemotherapy in locally advanced head and neck cancers : Secondary results of two European randomized phase III trials (ARO 95-06, SAKK 10/94). Strahlenther Onkol. 2016 Aug;192(8):552-60. doi: 10.1007/s00066-016-0999-3. Epub 2016 Jun 20. PMID 27323753
- [Result] Ghadjar P, Hayoz S, Zimmermann F, Bodis S, Kaul D, Badakhshi H, Bernier J, Studer G, Plasswilm L, Budach V, Aebersold DM; Swiss Group for Clinical Cancer Research (SAKK). Impact of weight loss on survival after chemoradiation for locally advanced head and neck cancer: secondary results of a randomized phase III trial (SAKK 10/94). Radiat Oncol. 2015 Jan 17;10:21. doi: 10.1186/s13014-014-0319-y. PMID 25679310
- [Result] Ghadjar P, Sun H, Zimmermann F, Bodis S, Bernier J, Studer G, Aebersold DM; Swiss Group for Clinical Cancer Research (SAKK). Physical examination during chemoradiation predicts outcome of locally advanced head and neck cancer. Secondary results of a randomized phase III trial (SAKK 10/94). Oral Oncol. 2013 Oct;49(10):1006-9. doi: 10.1016/j.oraloncology.2013.07.002. Epub 2013 Aug 3. PMID 23916716